CLINICAL TRIAL: NCT03830801
Title: Pilot Study for OCT Guided In Vivo Laser Capture Microdissection for Assessing the Prognosis of Barrett's Esophagus
Acronym: IVLCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-P001752; 5R01EB022077-02 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett Esophagus
Keywords: Barrett's Esophagus; EGD; Endoscopy; Biopsy; Tethered Capsule Endomicroscopy; OCT
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IVLCM tethered capsule for biopsies (Experimental): IVLCM tethered capsule for obtaining biopsies for genomic sequencing of BE for the assessment of EAC risk.
  Interventions: Device: IVLCM tethered capsule

INTERVENTIONS:
Device: IVLCM tethered capsule — Obtaining biopsies for genomic sequencing of BE for the assessment of EAC risk using IVLCM tethered capsule

SUMMARY:
The investigators have developed a new technology, termed in-vivo laser capture microdissection (IVLCM), that addresses the limitations of endoscopic biopsy for screening for BE and provides targeted genomic profiling of aberrant tissue for more precise prediction of EAC risk. The device is a tethered capsule endomicroscope (TCE) that implements optical coherence tomography (OCT) to grab 10-mm-resolution, cross-sectional microscopic images of the entire esophagus after the capsule is swallowed. This OCT-based TCE technology is used in unsedated patients to visualize images of BE and dysplastic BE. During the IVLCM procedure, TCE images of abnormal BE tissue are identified in real time and selectively adhered onto the device. When the capsule is removed from the patient, these tissues, targeted based on their abnormal OCT morphology, are sent for genomic analysis. By enabling the precise isolation of aberrant esophageal tissues using a swallowable capsule, this technology has the potential to solve the major problems that currently prohibit adequate BE screening and prevention of Esophageal Adenocarcinoma EAC.

DETAILED DESCRIPTION:
In Vivo Laser Capture Microdissection (IVLCM). The IVLCM tethered capsule is identical to those used in current approved OCT TCE studies.The capsule is swallowed by the patient and then, in real time, a region for tissue capture, is identified on the images. When a targeted site is identified, a capture laser (1450 nm, 0.8 W, 1 second exposure; within the range of the previously approved OCT-TCE tissue marking study) irradiates this area in the patient, heating the water in the tissue and transforming it to steam. The accumulated water steam overcomes the tissue matrix's adhesion force, ejecting a small amount of tissue and integrating it with the capsule's external shell. This process may then be repeated to collect multiple samples. After the device is pulled out from the patient, the captured tissues can be extracted for genomic analysis. Ex vivo animal tissue studies have shown that capture laser does not damage DNA/RNA; high quality whole genome information can be obtained.

In this IVLCM study, the investigators are using a 1450 nm laser to capture tissue that was previously approved to make cautery "marks" in the esophagus. The IVLCM capture laser's specifications are the same as those of the marking laser and the power will be within the IRB approved power range (0.82 W 1s). Prior to testing laser marking in humans, the investigators first demonstrated the safety of laser marking in animals in vivo. Histological assessment showed that the cautery marks did not penetrate through the submucosa and the vast majority of the effects were limited to the epithelium, lamina propria, and muscularis mucosa layers. The extent of thermal damage was comparable to conventional biopsies in standard of care endoscopic biopsy procedures. After this animal study, the investigators conducted a pilot study in humans in which over 30 marks were made in 22 enrolled subjects without any adverse events or safety concerns. In addition to these balloon studies, the investigators are currently conducting a TCE marking study. So far, the investigators have imaged and marked 13 subjects through a capsule without any adverse effects or safety concerns.

Thirty (N=30) subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a current or prior diagnosis of Barrett's Esophagus
* Participants must be over the age of 18.
* Participants must be able to give informed consent.

Exclusion Criteria:

* Pregnant women.
* Participants who are on anti-platelet medications or anti-coagulation medications, and NSAIDS at the time of procedure.
* Participants with a history of hemostasis disorders.
* Participants with esophageal strictures, resulting in a luminal diameter smaller than the diameter of the capsule.
* Participants with a know history of esophageal varices
* Participants above 80 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants from which we will be able to collect biopsy samples using IVLCM technique | 5 months
  We will measure the number of subjects from which we will be able to collect biopsy samples using IVLCM technique

CONTACTS AND LOCATIONS:
Overall Officials: Gary Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No